CLINICAL TRIAL: NCT07333469
Title: A Phase I/IIa Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Clinical Efficacy of HX111 in Patients With Advanced Solid Tumor and Lymphoma
Brief Title: A Clinical Study of HX111 in Patients With Advanced Solid Tumor and Lymphoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hanx Biopharmaceuticals (Wuhan) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX111-I-01
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor and Lymphoma
Keywords: Phase I/IIa
MeSH Terms: conditions — Lymphoma | interventions — Injections

STUDY DESIGN:
Intervention Model Description: The study will consist of a Phase I dose-escalation and Phase IIa dose-expansion component. Phase I dose-escalation phase will establish the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D),and evaluate the preliminary antitumor activity of HX111.
  Phase I dose-escalation phase Eligible patients with advanced solid tumors and lymphoma will be enrolled. The total sample size is up to 54 patients enrolled for DLT evaluable population. Dose-limiting toxicities (DLTs) will be assessed from the first dose of study treatment (Day 1) until 21 days later (Day 22).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention arm (Experimental): HX111 for injection
  Interventions: Drug: HX111 for injection

INTERVENTIONS:
Drug: HX111 for injection — HX111, 0.5-2.5mg/kg, once every 3 weeks

SUMMARY:
The study will consist of a Phase I dose-escalation and Phase IIa dose-expansion component. Phase I dose-escalation phase will establish the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D),and evaluate the preliminary antitumor activity of HX111.

DETAILED DESCRIPTION:
Phase I dose-escalation phase Eligible patients with advanced solid tumors and lymphoma will be enrolled. The total sample size is up to 54 patients enrolled for DLT evaluable population. Dose-limiting toxicities (DLTs) will be assessed from the first dose of study treatment (Day 1) until 21 days later (Day 22).

The dose escalation will be guided by Bayesian optimal interval (BOIN) design. The target toxicity rate ϕ is 0.3, The alternative hypothesis toxicity rates are ϕ_1=0.6ϕ and ϕ_2=1.4ϕ, respectively. The posterior probability threshold for dose elimination is 0.95. The maximum number of evaluable subjects per dose group is 9. Dose escalation will continue until one of the following criteria is met

ELIGIBILITY:
Inclusion Criteria:

* 1. Able to understand and voluntarily sign the Informed Consent Form (ICF); 2. Male or female subject aged 18 to 70 years, inclusive. 3. Eastern Cooperative Oncology Group performance status of 0 to 1. 4. Life expectancy of ≥3 months; 5. Histologically confirmed advanced solid tumors (including sarcomas, head and neck squamous carcinoma, cervical cancer, breast cancer, etc.,) or advanced lymphomas (including peripheral T-cell lymphoma-not otherwise specified, Angioimmunoblastic T-cell Lymphoma, Extranodal Natural Killer/T-cell Lymphoma (nasal type), adult T-cell lymphoma/leukemia, Anaplastic Large Cell Lymphoma, and other EBV+ lymphomas) that is refractory/relapsed to standard therapies, or for which no effective standard therapy , or or for which the subject refuses standard treatment is available,.

  6. For advanced solid tumors At least one measurable lesion per RECIST v1.1; 7. For patients with lymphoma:

  • Lymphoma diagnosed according to the 2022 WHO Classification, 5th Edition, and meeting the definition of relapsed/refractory disease.

  • At least one measurable lesion according to the Lugano criteria within 4 weeks prior to the first dose; Measurable lesion: Lymph node with the longest diameter >15 mm, extranodal lesions >10 mm; Lesions previously treated with radiotherapy or other local therapies are considered measurable if disease progression has been documented and they meet the definition of measurable lesions.

Inclusion Criteria

1. Able to understand and voluntarily sign the Informed Consent Form (ICF);
2. Male or female subject aged 18 to 70 years, inclusive.
3. Eastern Cooperative Oncology Group performance status of 0 to 1.
4. Life expectancy of ≥3 months;
5. Histologically confirmed advanced solid tumors (including sarcomas, head and neck squamous carcinoma, cervical cancer, breast cancer, etc.,) or advanced lymphomas (including peripheral T-cell lymphoma-not otherwise specified, Angioimmunoblastic T-cell Lymphoma, Extranodal Natural Killer/T-cell Lymphoma (nasal type), adult T-cell lymphoma/leukemia, Anaplastic Large Cell Lymphoma, and other EBV+ lymphomas) that is refractory/relapsed to standard therapies, or for which no effective standard therapy , or or for which the subject refuses standard treatment is available,.
6. For advanced solid tumors At least one measurable lesion per RECIST v1.1;
7. For patients with lymphoma:

   • Lymphoma diagnosed according to the 2022 WHO Classification, 5th Edition, and meeting the definition of relapsed/refractory disease.

   • At least one measurable lesion according to the Lugano criteria within 4 weeks prior to the first dose; Measurable lesion: Lymph node with the longest diameter >15 mm, extranodal lesions >10 mm; Lesions previously treated with radiotherapy or other local therapies are considered measurable if disease progression has been documented and they meet the definition of measurable lesions.
8. Adequate organ function, as indicated by the following laboratory values, within 7 days before first dose (unless specified):

   Hematology (use of hematopoietic growth factors and transfusions not allowed within 14 days prior to the start of the first study treatment) • Absolute neutrophil count (ANC) ≥1.5 × 109/L; for those with bone marrow involvement, ANC ≥1.0 × 109/L Solid tumor

   • Hemoglobin ≥100 g/L

   • Platelet count ≥100 × 109/L lymphoma

   • Hemoglobin (HB) ≥90 g/L; for those with bone marrow involvement, HB ≥80 g/L;

   • Platelet count ≥75×109/L (without bone marrow involvement), platelet count ≥50.0×109/L (with bone marrow or splenic involvement)； Hepatic：

   • Serum total bilirubin ≤1.5×upper limit of normal (ULN); or for patients with total bilirubin levels >1.5ULN but direct bilirubin ≤ULN

   • Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN (for subjects with liver metastases, ALT and AST ≤5×ULN) Renal：

   • Serum creatinine ≤1.5×ULN Coagulation function ( within 14 days before first dose)：

   • Prothrombin time/International Normalized Ratio ≤1.5×ULN or activated partial thromboplastin time ≤1.5×ULN (for subjects receiving anticoagulants, the prothrombin time or activated partial thromboplastin time must be within the normal range for their anticoagulant regimen)。 Echocardiogram ( within 28 days before first dose)：
   * LVEF≥50%
9. Male subjects: Must agree to use the contraception methods recommended in Appendix 5 during the treatment period and for at least 12 months after the last dose of the study treatment.

Female subjects: Contraception; or not having reproductive potential as defined in Appendix 5; or if of reproductive potential, must agree to use effective contraception during the study treatment period and for at least 12 months after the last dose of study treatment. Female subjects of reproductive potential are required to have a negative pregnancy test within 14 days before administration of the study drug.

Exclusion Criteria:

* 1. Prior malignancy active within the previous 2 years except for the tumor for which a subject is enrolled in the study and locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast.

Known allergic reactions to prior recombinant humanized anti-OX40 monoclonal antibody drugs or their components.

2. Received any anti-tumor treatment (chemotherapy, radiotherapy, study drugs including small molecule inhibitors, endocrine therapy, immunotherapy, etc.) within 4 weeks or 5 half-lives of that treatment (whichever is shorter) prior to the first dose of study treatment .

3. Received any investigational anti-tumor treatment within 4 weeks prior to the first dose of study treatment 4. History of Grade ≥2 peripheral neuropathy 5. Toxicities from prior anti-tumor treatments have resolved to ≤Grade 1 or to baseline, with the exception of alopecia and Grade 2 hypothyroidism that can be managed with hormone replacement therapy.

6. Any subject known to be positive for human immunodeficiency virus, or active hepatitis B virus or hepatitis C virus infection.

7. Female subject who is pregnant or lactating. 8. Subjects with a history of or presently experiencing an active autoimmune disease (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulitis, etc.) within 2 years of initiating study drug, or those who are at high risk of relapse (e.g., receiving an immunosuppressive treatment for an organ transplant); however, subjects with the following are allowed to enroll:

* Type I diabetes that is stable after a fixed dose of insulin or other hypoglycemic
* Only requiring hormone replacement therapy for autoimmune hypothyroidism
* Skin disease that does not require systemic treatment such as eczema, rash that accounts for <10% of the body surface, psoriasis without ophthalmic symptoms.

  9. Subjects who have undergone any major surgery (excluding diagnostic surgery) within 4 weeks prior to the first study treatment, and/or subjects who may require major surgery during the study period including the screening period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2028-01-19 (Estimated); Study Completion 2030-01-19 (Estimated)

PRIMARY OUTCOMES:
DLTs | 21 days
  rate of DLTs

SECONDARY OUTCOMES:
ORR | 24 months
  rate of response

IPD SHARING:
Plan to Share IPD: No